CLINICAL TRIAL: NCT02708901
Title: Gut to Brain Interaction in Autism. Role of Probiotics on Clinical, Biochemical and Neurophysiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Ministry of Health, Italy (Other Government); Istituto di Fisiologia Clinica CNR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR-2011-02348280
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2017-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Probiotic Vivomixx®; Gastrointestinal Symptoms; Gut-Brain Axis; Endophenotypes
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized double blind study of dietary supplement compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GI Vivomixx® (Active Comparator): 25 children with GI symptoms
  Interventions: Dietary Supplement: Vivomixx®
- GI Placebo (Placebo Comparator): 25 children with GI symptoms
  Interventions: Dietary Supplement: Placebo
- NGI Vivomixx® (Active Comparator): 25 children without GI symptoms
  Interventions: Dietary Supplement: Vivomixx®
- NGI placebo (Placebo Comparator): 25 children without GI symptoms
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx® — Two packets (900 billions bacteria) per os (P.O.) daily x 1 month and one packet (450 billions bacteria) P.O. daily x 5 months
  Arms: GI Vivomixx®; NGI Vivomixx®
Dietary Supplement: Placebo — Two packets (4,4 grams of maltose and silicon dioxide x 2) P.O. daily x 1 month and one packet (4,4 grams of maltose and silicon dioxide) P.O. daily x 5 months
  Arms: GI Placebo; NGI placebo

SUMMARY:
The purpose of this study is to assess the effects of a 6-months supplementation with probiotic Vivomixx® on inflammatory and gastrointestinal (GI) biomarkers, gastrointestinal disturbances, behavioral and developmental profiles, and neurophysiological features in preschoolers with Autism Spectrum Disorders (ASD) with or without GI symptoms.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are most likely multifactorial diseases in which the combination of genetic and environmental factors might have a role in the expression of the phenotype. A high incidence of gastrointestinal (GI) symptoms is reported in ASD. GI disturbances and altered gut microflora could make a child with a genetic predisposition for ASD more prone to express the ASD phenotype or increase the severity of his behavioral symptoms. The exploitation of strategies which can reduce the gut production and absorption of toxins or restore normal gut microbiota, such as probiotics may represent a non-pharmacological option in the treatment of GI disturbances in ASD. The aim of this study is to determine effects of probiotics supplementation with Vivomixx® in ASD children on specific GI symptoms, ASD core deficits, cognitive and language development, on inflammatory and gastrointestinal (GI) biomarkers and on Quantitative Electroencephalographic measures (QEEG). Vivomixx® is a probiotic mixture of 8 probiotic strains (Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, Lactobacillus bulgaricus and Streptococcus thermophilus). An additional aim of the study is to determine the environmental exposure to phthalates (chemical pollutant) in ASD children, and the possible effects of probiotic supplementation on their urinary concentrations. A group of 100 unselected preschoolers with ASD will be classified as belonging to the Gastro Intestinal (GI) group or to the Not Gastro Intestinal (NGI) group on the basis of the presence of significant GI symptoms at GI severity Index. Subjects belonging to the two groups (GI and NGI) will be blind randomized 1:1 to regular diet with probiotic Vivomixx® or with placebo for 6 months. All the participants will be assessed at the baseline, after three months and after six months from the baseline in order to evaluate the possible changes in GI symptoms, in ASD symptomatology, in other affective and behavioral comorbid symptoms, in plasmatic, urinary and fecal biomarkers related to abnormal intestinal function and in the electrophysiological patterns. The effects of treatments with probiotics on children with ASD need to be confirmed by rigorous controlled trials. Aiming to examine the impact of this treatment not only on clinical but also on neurophysiological patterns this trial sets out to provide new insights into the gut-brain connection in autism. Moreover, this study's results could add new data on the relationship between the presence of phthalates, clinical features and neurophysiological patterns in ASD.

ELIGIBILITY:
Inclusion Criteria:

* age-range: 18-72 months
* ASD diagnosis according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria

Exclusion Criteria:

* brain anomalies detected by Magnetic Resonance Imaging (MRI)
* neurological syndromes or focal neurological signs
* anamnesis of birth asphyxia, severe premature birth (≤ 28 gestational weeks) or perinatal injuries
* epilepsy
* significant sensory impairment
* diagnosis of organic GI Disorder (i.e. gastroesophageal reflux, food allergies, Inflammatory Bowel Disease)
* diagnosis of Coeliac Disease
* special diet (i.e. gluten-free diet, casein-free diet, high-protein diet, ketogenic diet)

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Changes in severity level of ASD symptomatology | 6 months
  Delta of scores at Autism Diagnostic Observation Schedule-2

SECONDARY OUTCOMES:
Changes in GI symptomatology | 3 months and 6 months
  Delta of scores at GI Severity Index
Changes in Electroencephalogram (EEG) power | 6 months
  Registration with a 128-channels digital EEG: power will be assessed within each frequency band
Changes in EEG coherence | 6 months
  Registration with a 128-channels digital EEG: coherence will be assessed within each frequency band
Changes in EEG asymmetry | 6 months
  Registration with a 128-channels digital EEG: asymmetry will be assessed within each frequency band
Changes in levels of serum Lipopolysaccharide | 6 months
  Delta of values of serum Lipopolysaccharide
Changes in levels of serum Leptin | 6 months
  Delta of values of serum Leptin
Changes in levels of serum Resistin | 6 months
  Delta of values of serum Resistin
Changes in levels of serum Tumor Necrosis Factor - alfa | 6 months
  Delta of values of serum Tumor Necrosis Factor - alfa
Changes in levels of serum Interleukin-6 (IL-6) | 6 months
  Delta of values of serum Interleukin-6 (IL-6)
Changes in levels of serum Plasminogen Activator Inhibitor-1 (PAI-1) | 6 months
  Delta of values of serum Plasminogen Activator Inhibitor-1 (PAI-1)
Changes in levels of fecal calprotectin | 3 months and 6 months
  Delta of values of fecal calprotectin
Changes in global ASD symptomatology assessed by Childhood Autism Rating Scale | 6 months
  Delta of scores at Childhood Autism Rating Scale
Changes in ASD symptomatology: repetitive behaviors | 3 months and 6 months
  Delta of scores at Repetitive Behavior Scale
Changes in ASD symptomatology: sensory profiles | 3 months and 6 months
  Delta of scores at Sensory Profile
Changes in global ASD symptomatology assessed by Social Communication Questionnaire | 3 months and 6 months
  Delta of scores at Social Communication Questionnaire
Changes in Developmental Quotient | 6 months
  Delta of score at Griffiths Mental Developmental Scale
Changes in Adaptive Functioning | 6 months
  Delta of scores at Vineland Adaptive Behavior Scale-II
Changes in Behavioral Profiles | 3 months and 6 months
  Delta of scores at Child Behavior Checklist 1.5-5
Changes in Parental Stress | 3 months and 6 months
  Delta of scores at Parenting Stress Index

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Santocchi, MD, PhD, Principal Investigator — IRCCS Stella Maris Foundation
Locations (1):
- IRCCS Stella Maris Foundation, Calambrone, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fulceri F, Morelli M, Santocchi E, Cena H, Del Bianco T, Narzisi A, Calderoni S, Muratori F. Gastrointestinal symptoms and behavioral problems in preschoolers with Autism Spectrum Disorder. Dig Liver Dis. 2016 Mar;48(3):248-54. doi: 10.1016/j.dld.2015.11.026. Epub 2015 Dec 11. PMID 26748423
- [Background] Santocchi E, Guiducci L, Fulceri F, Billeci L, Buzzigoli E, Apicella F, Calderoni S, Grossi E, Morales MA, Muratori F. Gut to brain interaction in Autism Spectrum Disorders: a randomized controlled trial on the role of probiotics on clinical, biochemical and neurophysiological parameters. BMC Psychiatry. 2016 Jun 4;16:183. doi: 10.1186/s12888-016-0887-5. PMID 27260271
- [Background] Calderoni S, Santocchi E, Del Bianco T, Brunori E, Caponi L, Paolicchi A, Fulceri F, Prosperi M, Narzisi A, Cosenza A, Tancredi R, Muratori F. Serological screening for Celiac Disease in 382 pre-schoolers with Autism Spectrum Disorder. Ital J Pediatr. 2016 Nov 16;42(1):98. doi: 10.1186/s13052-016-0308-x. PMID 27852289
- [Background] Prosperi M, Santocchi E, Balboni G, Narzisi A, Bozza M, Fulceri F, Apicella F, Igliozzi R, Cosenza A, Tancredi R, Calderoni S, Muratori F. Behavioral Phenotype of ASD Preschoolers with Gastrointestinal Symptoms or Food Selectivity. J Autism Dev Disord. 2017 Nov;47(11):3574-3588. doi: 10.1007/s10803-017-3271-5. PMID 28861653
- [Derived] Santocchi E, Guiducci L, Prosperi M, Calderoni S, Gaggini M, Apicella F, Tancredi R, Billeci L, Mastromarino P, Grossi E, Gastaldelli A, Morales MA, Muratori F. Effects of Probiotic Supplementation on Gastrointestinal, Sensory and Core Symptoms in Autism Spectrum Disorders: A Randomized Controlled Trial. Front Psychiatry. 2020 Sep 25;11:550593. doi: 10.3389/fpsyt.2020.550593. eCollection 2020. PMID 33101079